CLINICAL TRIAL: NCT03471975
Title: Comparison of Training Effect for Tracheal Intubation Following Training With McGrath Video Laryngoscope as Direct Laryngoscope Versus Training With McGrath Video Laryngoscope as Video Laryngoscope
Brief Title: Learning Direct Laryngoscopy Using a McGrath Video Laryngoscope as Direct Versus Indirect Laryngoscope
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ajou University School of Medicine (Other)
Responsible Party: Principal Investigator, Jihoon Hwang, MD, Clinical Assistant Professor, Ajou University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: AJIRB-SBR-OBS-17-507
Record Dates: First submitted 2018-03-09; First posted 2018-03-21 (Actual); Results first posted 2019-08-19 (Actual); Last update posted 2019-08-19 (Actual); Status verified 2019-07

CONDITIONS: Airway Management; Endotracheal Intubation; Medical Education
Keywords: Video laryngoscopy

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- direct laryngoscope (Active Comparator): teaching tracheal intubation using McGrath video laryngoscope as direct laryngoscope. Only trainer can see the monitor.
  Interventions: Procedure: direct laryngoscope
- video laryngoscope (Active Comparator): teaching tracheal intubation using McGrath video laryngoscope using video function.
  Trainer and Trainee both see the monitor.
  Interventions: Procedure: video laryngoscope

INTERVENTIONS:
Procedure: direct laryngoscope — the trainee use McGrath video laryngoscope as direct laryngoscope the trainee is not allowed to watch the screen.
  Arms: direct laryngoscope
Procedure: video laryngoscope — the trainee use McGrath video laryngoscope both trainee and trainer can watch the screen.
  Arms: video laryngoscope

SUMMARY:
prospective randomised trial to compare the teaching effect for tracheal intubation following training with McGrath video laryngoscope as direct laryngoscope versus training with McGrath video laryngoscope as video laryngoscope

DETAILED DESCRIPTION:
Tracheal intubation using direct laryngoscopy is very important technique in clinical medicine. But the training for intubation is not very easy because laryngoscopic view is difficult to share between trainee and trainer.

Recently there have been reported that tracheal intubation training using video laryngoscopy have some advantages and showed more success rate.

McGrath Video laryngoscopy can be used as either video laryngoscopy or direct laryngoscopy. Therefore when McGrath is used as intubation training tool, the trainer can monitor and educate the procedure while the trainee perform tracheal intubation.

The aim of this study is comparing the teaching effect for tracheal intubation following training with McGrath video laryngoscope as direct laryngoscope versus training with McGrath video laryngoscope as video laryngoscope

ELIGIBILITY:
Inclusion Criteria:

* medical students who has never experienced intubation

Exclusion Criteria:

* A person who has previously experienced intubation with Manikin or patients.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2018-03-12 (Actual); Primary Completion 2018-07-09 (Actual); Study Completion 2018-07-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jihoon Hwang, MD, Principal Investigator — Clinical Assistant Professor
Locations (1):
- Ajou University School of Medicine, Suwon, Gyeonggi-do, South Korea

REFERENCES:
- [Derived] Yi IK, Hwang J, Min SK, Lim GM, Chae YJ. Comparison of learning direct laryngoscopy using a McGrath videolaryngoscope as a direct versus indirect laryngoscope: a randomized controlled trial. J Int Med Res. 2021 May;49(5):3000605211016740. doi: 10.1177/03000605211016740. PMID 34024186

RESULTS

PARTICIPANT FLOW:
Groups:
- Video Laryngoscope: teaching tracheal intubation using McGrath video laryngoscope using video function.
  Trainer and Trainee both see the monitor.
  video laryngoscope: the trainee use McGrath video laryngoscope both trainee and trainer can watch the screen.
Period: Overall Study
Arm/Group | Direct Laryngoscope | Video Laryngoscope
Started | 17 | 20
Completed | 17 | 20
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Direct Laryngoscope | Video Laryngoscope | Total
Number analyzed (Participants) | 17 | 20 | 37
Age, Continuous [Mean (Standard Deviation); unit: years] | 24.8 (1.5) | 24.7 (1.5) | 24.8 (1.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 9 | 16
  Male | 10 | 11 | 21
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 17 | 20 | 37
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Intubation Success Rate
Description: tracheal intubation success rate using direct laryngoscope on manikin
Time Frame: up to 10 minutes
Measure: Count of Participants; unit: Participants
Arm/Group | Direct Laryngoscope | Video Laryngoscope
Number analyzed (Participants) | 17 | 20
Participants | 14 | 14

2. Primary Outcome: Time to Intubation
Description: Time from device passing the mouth until confirmation of tracheal intubation
Time Frame: up to 10 minutes
Measure: Mean (Full Range); unit: second
Arm/Group | Direct Laryngoscope | Video Laryngoscope
Number analyzed (Participants) | 17 | 20
second | 54.6 [22 to 100] | 56.8 [25 to 100]

ADVERSE EVENTS:
Time Frame: 5 months
Arm/Group | Direct Laryngoscope | Video Laryngoscope
All-Cause Mortality (participants affected / at risk) | 0/17 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/17 | 0/20
Other Adverse Events (participants affected / at risk) | 0/17 | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-03-01): https://cdn.clinicaltrials.gov/large-docs/75/NCT03471975/Prot_SAP_000.pdf